CLINICAL TRIAL: NCT00264784
Title: The Epidemiology of Group A Streptococcal Infections in Fiji (Fiji GrASP) - Part 5: Establishing Natural Age-Related Titers of Antibodies to the J8 Group A Streptococcal Epitope in Fiji
Brief Title: GAS Epi Study to Measure Age-Related Antibody Titers to J8 Vaccine
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Other Study IDs: 05-0081
Record Dates: First submitted 2005-12-09; First posted 2005-12-13 (Estimated); Last update posted 2007-12-28 (Estimated); Status verified 2007-10

CONDITIONS: Streptococcus Group A
Keywords: Streptococcus, Group A, Fiji, epidemiology

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
The purpose of this ongoing study (Part V) is to evaluate the cause, distribution, control, and results of group A streptococcus infections (GAS) in Fiji. Patients of all ages presenting to the Colonial War Memorial Hospital, Suva, Fiji and patients donating blood to the Colonial War Memorial Hospital, Suva, Fiji may participate. Subject duration is less than one day. This study may help to develop a vaccine that will prevent group A streptococcal infections.

DETAILED DESCRIPTION:
Most group A streptococcus (GAS) disease occurs in childhood and the premise of this study is that with increasing age there is apparent clinical protection from GAS disease which is due to the acquisition of protective antibodies. The study therefore seeks to test the hypothesis that titers of anti-J8 antibodies will increase with increasing age. This study is part 5 of a series including Division of Microbiology and Infectious Diseases (DMID) protocols 05-0082, 05-0117, 05-0118, and 06-0081. Three hundred patients will be selected in 6 age groups with 50 patients in each group: 0-4 years of age, 5-14 years of age, 15-24 years of age, 25-34 years of age, 35-49 years of age, over 50 years of age. Participants will be recruited through the Colonial War Memorial (CWM) Hospital in Suva. Patients in the hospital who are having blood taken for reasons other than GAS disease will be approached and asked to participate in the study. These patients will include people who are donating blood to the blood collection service for CWM Hospital. In addition, it will include patients going to the operating room or patients having blood taken as an outpatient by the pathology blood collection service. Once informed consent is obtained, blood will be collected in a serum separator blood tube. The volume of blood required for age groups will vary: 3ml whole blood for those aged <5 years, 5 mls for those aged 5-14 years, 7.5 mls for those aged greater than 14 years. Participants will be excluded if they have a history of serious GAS disease including acute rheumatic fever, acute post streptococcal glomerulonephritis, invasive disease, or rheumatic heart disease, or if they have had a sore throat or skin sores within the past 14 days. These participants will be excluded because it is not known if J8 titres may correlate with prior serious GAS diseases or if there is an acute J8 antibody response to recent GAS infection, and we are aiming to understand background titres of J8 antibodies in this population. In addition, these illnesses will affect the value of antistreptolysin O titre (ASOT) and anti-DNase-B to establish the upper limits of normal values. After blood is centrifuged it will be divided. Aliquots will be prepared for measurement of ASOT and anti-DNase B titers. Further aliquots will be stored in the laboratory and sent to Queensland Institute of Medical Research in batch for measurement of J8 antibodies.

ELIGIBILITY:
Inclusion Criteria:

Individuals of any age who are inpatients or outpatients at Colonial War Memorial Hospital and provide informed consent.

Exclusion Criteria:

Patients will be excluded from participating in the study if they have a history of acute rheumatic fever, acute post streptococcal glomerulonephritis, rheumatic heart disease, or invasive Group A Streptococcus disease or have had a sore throat or skin sores within the past 14 days as determined by self report, or if they have a current febrile illness (>38.0 degrees Celsius).

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 300
Dates: Start 2005-12; Study Completion 2006-05

CONTACTS AND LOCATIONS:
Locations (1):
- Colonial War Memorial Hospital, Suva, Fiji